CLINICAL TRIAL: NCT06147921
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Verasone™ Administered by Sinonasal Irrigation in Healthy Participants
Brief Title: Phase 1, SAD/MAD of Verasone™ Administered by Sinonasal Irrigation in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Diceros Therapeutics (Industry)
Collaborators: Diceros Therapeutics Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VER-001
Record Dates: First submitted 2023-11-02; First posted 2023-11-28 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose (SAD), Single Dose Active Components PK Crossover, Multiple Ascending Dose (MAD)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- SAD Dose Level 1 (Experimental): Sinonasal irrigation of lowest dose Verasone vs placebo
  Interventions: Drug: Verasone
- SAD Dose Level 2 (Experimental): Sinonasal irrigation of second lowest dose Verasone vs placebo
  Interventions: Drug: Verasone
- SAD Dose Level 3 (Experimental): Sinonasal irrigation of third lowest dose Verasone vs placebo
  Interventions: Drug: Verasone
- SAD Dose Level 4 (Experimental): Sinonasal irrigation of highest dose Verasone vs placebo
  Interventions: Drug: Verasone
- Crossover Component (Active Comparator): Each active component from the highest well tolerated dose of Verasone will be administered via sinonasal irrigation alone in a within subject crossover to compare plasma drug levels to that seen when dosed with Verasone.
  Interventions: Drug: Verasone
- MAD Dose Level 1 (Experimental): The next to highest well tolerated dose of Verasone in the SAD study will be compared to one of the active components in Verasone and to placebo in a 5 day b.i.d. dosing regimen
  Interventions: Drug: Verasone
- MAD Dose Level 2 (Experimental): The highest well tolerated of Verasone in the SAD study will be compared to one of the active components in Verasone and to placebo in a 5 day b.i.d. dosing regimen.
  Interventions: Drug: Verasone

INTERVENTIONS:
Drug: Verasone — Administered by sinonasal irrigation.

SUMMARY:
Verasone™ is an aqueous suspension of the combination of two marketed drugs to be dosed by sinonasal irrigation in the treatment of Chronic Rhinosinusitis (CRS). This Phase 1 first-in-human study will assess the safety, tolerability, and pharmacokinetics (PK) of single and multiple ascending doses of Verasone versus placebo in healthy normal participants and will evaluate the PK profiles of the Verasone active components administered individually vs in combination.

ELIGIBILITY:
Main Inclusion Criteria:

1. In good general health based on medical history, physical examination, vital signs, ECG, laboratory parameters, and other relevant tests
2. Able to perform study procedures, including self-administration of sinonasal irrigation of 60 mL in each nostril
3. Able and willing to attend the necessary visits to the study site.

   Additional inclusion criteria for Part B:
4. Participant met all eligibility criteria for Part A, completed Part A with no major protocol deviations, and all Part A safety and PK assessments were completed, in the opinion of the PI.
5. Participant did not experience local toxicity AEs or anterior rhinoscopy findings during Part A.

Main Exclusion Criteria:

1. History of allergy, hypersensitivity, or contraindication to corticosteroids or calcium channel blockers.
2. History of severe allergic or anaphylactic reactions or sensitivity to the IP or its constituents.
3. Any clinical obstruction of the nasal cavities that would reduce access for topical irrigations
4. Nasal candidiasis, nasal mucosal ulceration, thinning or eroded nasal septum, or nasal septum perforation.
5. History or clinical evidence of CRS, fungal rhinosinusitis, or rhinitis medicamentosa at any time, or any active allergic rhinitis, acute sinusitis, or upper respiratory infection within 4 weeks prior to Screening.
6. Ongoing nasal congestion at Screening or Day -1 (Nasal Congestion Score > 0).
7. Inability to have anterior rhinoscopy nasal examination (Parts A and B only) or endoscopic nasal cavity examination (Part C only).
8. More than 1 episode of epistaxis.
9. History of or planned sinus or intranasal surgery.
10. Use of immunomodulating drugs, except glucocorticoids, within 90 days prior to Screening or intent to use these drugs during the study.
11. Exposure to any glucocorticoid treatment via any route (nasal, topical, inhaled, oral, intravenous, etc.) within 1 month prior to Screening.
12. Received biologic therapy/systemic immunosuppressant to treat inflammatory or autoimmune disease.
13. Oral steroid-dependent or monoclonal antibody-dependent (eg, omalizumab, mepolizumab, dupilumab) condition.
14. Use of potent cytochrome P450 3A4 (CYP3A4) inhibitor(s) or inducer(s) within 14 days prior to Screening.
15. Known history of HPA axial dysfunction, or previous pituitary or adrenal surgery.
16. History or diagnosis of eustachian tube dysfunction, recurrent otitis media.
17. Any history or ongoing clinically significant cardiac disease.
18. Abnormal vital signs or ECG findings.
19. History or current diagnosis of any form of glaucoma or ocular hypertension.
20. A history of cancer, HIV, or other immunodeficiency, or immune system-mediated disorder.
21. History of insulin-dependent diabetes mellitus.
22. History of any clinically significant hepatic or renal disease.
23. Clinically significant abnormal laboratory parameters at Screening.
24. Any underlying physical or psychological medical condition.
25. A recent clinically significant history of drug or alcohol use, abuse, or dependence.
26. Positive screen for drugs of abuse or alcohol at Screening or Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Part A: Single Ascending Dose (SAD) | 1 week
  The proportion of subjects with Adverse Events at each dose level
Part B: Single Dose Component Crossover | 3 weeks
  Plasma drug levels of Verasone's components
Part C: Multiple Ascending Dose (MAD) | 2 weeks
  The proportion of subjects with Adverse Events at each dose level

SECONDARY OUTCOMES:
To assess the volume of retained fluid and amount of mucosal absorption in the sinonasal system immediately following single dose Verasone vs placebo administered by sinonasal irrigation in healthy participants. | 30 min
  To assess the volume of fluid retained in the sinonasal system following dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Data will be summarised as an aggregate per cohort.